CLINICAL TRIAL: NCT05673642
Title: Effect of Myofascial Release Therapy Applied to Selective Muscles on Mobility and Function in Patients With Temporomandibular Dysfunction: A Randomized Controlled Trial
Brief Title: Myofascial Release Therapy for TMD Pain: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ebru Senel T, PhD student., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-6577
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Temporomandibular Joint Disorder; Low Back Pain; Myofascial Release
Keywords: TMJ Disorder, Myofascial Release, Low back pain
MeSH Terms: conditions — Temporomandibular Joint Disorders; Low Back Pain

STUDY DESIGN:
Intervention Model Description: A parallel-group randomized controlled trial with three distinct arms.
Masking Description: This study was conducted as a single-blind randomized controlled trial, where participants were unaware of their group assignments. The care provider, investigator, and outcome assessor were also blinded to the group allocation to minimize assessment bias. The randomization process was conducted independently to ensure allocation concealment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Working group (Experimental): A total of 10 sessions will be applied myofascial release technique for 4 weeks, 3 times a week for the first 2 weeks, and 2 times a week for the next 2 weeks. Evaluations will be made at the beginning of the study and at the end of 4 weeks
  Interventions: Other: Myofascial Release Techniques
- Exercise group (Experimental): The stretching exercises that we planned to give to the exercise group were planned for the muscles to which we will apply myofascial technique. Evaluations will be made at the beginning of the study and at the end of 4 weeks
  Interventions: Other: Myofascial Release Techniques
- Control group (Experimental): No application will be made to the control group. Evaluations will be made at the beginning of the study and at the end of 4 weeks
  Interventions: Other: Myofascial Release Techniques

INTERVENTIONS:
Other: Myofascial Release Techniques — Myofascial Release Technique (MFR), which we will apply to the muscles we choose related to the facial system connection
  Other Names: Myofascial Exercise

SUMMARY:
We aim to compare the effectiveness of MFR and exercise therapy on mobility and function by investigating the effectiveness of the Myofascial Release Technique (MFR), which we will apply to the muscles we choose related to the facial system connection in participants with temporomandibular dysfunction (TMD) and low back pain.

DETAILED DESCRIPTION:
We aim to compare the effectiveness of MFR and exercise therapy on mobility and function by investigating the effectiveness of the Myofascial Release Technique (MFR), which we will apply to the muscles we choose related to the facial system connection in participants with temporomandibular dysfunction (TMD) and low back pain.

Method and Material Working group (Group A): Myofascial release technique will be applied. A total of 10 sessions will be applied for 4 weeks, 3 times a week for the first 2 weeks, and 2 times a week for the next 2 weeks.

Exercise group (Group B): The stretching exercises that we planned to give to the exercise group were planned for the muscles to which we will apply myofascial technique.

• Control group (Group C): No application will be made to the control group. Evaluations will be made at the beginning of the study and at the end of 4 weeks. The evaluation parameters to be used are as follows; Oswestry Low Back Disability Survey, Algometer and Myotonometry.

Inclusion Criteria: Participants aged 18-50 years diagnosed with TMD,Persons with a score of 20% or more on the Oswestry waist index, and People with low back pain for more than 3 months,Persons with mechanical low back pain and lumbar disc herniation without neurological deficits will be included in the study.Persons with acute or chronic temporomandibular dysfunction will be included. Exclusion Criteria; Neurological problems,Presence of extruded and sequestered lumbar disc herniation,Cardiovascular symptoms and circulation problems,Infection,Fibromyalgia, Acute arthritis conditions,Those with spinal abnormalities,Fracture history, presence of dislocation / subluxation will be excluded

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-50 years diagnosed with TMD
* Persons with a score of 20% or more on the Oswestry waist index, and
* People with low back pain for more than 3 months
* Persons with mechanical low back pain and lumbar disc herniation without neurological deficits will be included in the study.
* Persons with acute or chronic temporomandibular dysfunction will be included

Exclusion Criteria:

* Neurological problems,
* Presence of extruded and sequestered lumbar disc herniation
* Cardiovascular symptoms and circulation problems,
* Infection,
* Fibromyalgia, Acute arthritis conditions
* Those with spinal abnormalities,
* Fracture history, presence of dislocation / subluxation will be excluded

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-06-24 (Actual)

PRIMARY OUTCOMES:
Algometer | 5 minute
  Pressure algometer will be used for temporomandibular joint pain. It will be applied to the lower masseter muscles and anterior temporalis muscles bilaterally on the lateral pole of the algometer and the average of three applications in each region will be taken.
Myotonometry | 10 minute
  It will be used to assess muscle tone differences. Myotonometry provides valid and reliable measurement of tissue stiffness. The measurement will be applied bilaterally to the masseter, temporalis, trapezius, erector spinal muscles, quadrates lumborum and TFL muscles.

SECONDARY OUTCOMES:
DC-TMD Evoluation | 10 minute
  The amount of mouth opening will be used to evaluate mandibular lateral shifts and mandibular protrusion.
Oswestry Low Back Disability Survey | 10 minute
  To be used to assess functional disability for the lower back

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Senel topaloglu, 1, Principal Investigator — Istanbul Medipol University Turkey Istanbul
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will publish my manuscript about this study, so researchers can access my individual participant data with this way.

REFERENCES:
- [Derived] Senel Topaloglu E, Budak M, Atilgan E, Kurt H. Effect of myofascial release therapy applied to selective muscles on mobility and function in patients with temporomandibular dysfunction and co-occurring chronic low back pain: A randomized controlled trial. Medicine (Baltimore). 2025 Aug 22;104(34):e44086. doi: 10.1097/MD.0000000000044086. PMID 40859519